CLINICAL TRIAL: NCT03800524
Title: Safety and Efficacy of Tauroursodeoxycholic (TUDCA) as add-on Treatment in Patients Affected by Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Safety and Efficacy of TUDCA as add-on Treatment in Patients Affected by ALS
Acronym: TUDCA-ALS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Humanitas Mirasole SpA (Other)
Collaborators: University of Ulm (Other); University of Sheffield (Other); University Hospital, Tours (Other); KU Leuven (Other); UMC Utrecht (Other); University of Dublin, Trinity College (Other); Bruschettini S.r.l. (Unknown); Istituto Superiore di Sanità (Other); Motor Neurone Disease Association (Unknown); European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H2020/755094/2017/IT-01; 2018-002722-22 (EudraCT Number); 755094 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2019-01-04; First posted 2019-01-11 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — ursodoxicoltaurine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tauroursodeoxycholic acid (TUDCA) (Experimental): * Tauroursodeoxycholic acid (TUDCA) 250 mg capsules
  * Doses: 4 capsules (1 g) twice daily 10-15 minutes after a meal
  * Mode of administration: orally
  * Duration: 18 months
  Interventions: Drug: Tauroursodeoxycholic Acid
- Reference therapy (Placebo Comparator): * Placebo capsules identical to active compound
  * Doses: 4 capsules (1 g) twice daily 10-15 minutes after a meal
  * Mode of administration: orally
  * Duration: 18 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tauroursodeoxycholic Acid — * Tauroursodeoxycholic acid (TUDCA) 250 mg capsules
  * Doses: 4 capsules (1 g) twice daily 10-15 minutes after a meal
  * Mode of administration: orally
  * Duration: 18 months
  Other Names: TUDCA; Tudcabil; Taurolite
  Arms: Tauroursodeoxycholic acid (TUDCA)
Drug: Placebo — * Placebo 250 mg capsules
  * Doses: 4 capsules (1 g) twice daily 10-15 minutes after a meal
  * Mode of administration: orally
  * Duration: 18 months
  Arms: Reference therapy

SUMMARY:
This is a Phase III, multi-centre, randomized, double-blind, placebo-controlled, parallel-group study to evaluate Safety and Efficacy of Tauroursodeoxycholic (TUDCA) as add-on Treatment in Patients Affected by Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
Enrolled patients will be randomized to one of two treatment arms: TUDCA or identical placebo by oral route. The randomization will be performed in a ratio one to one for the two arms.

TUDCA will be administered orally at the dose of 1 g twice daily (2 g daily) for 18 months. Patients will be taking also riluzole at the dose of 50 mg twice daily (100 mg daily).

Patient randomization will take place after a screening (lead-in) period of 12 weeks (3 months) with 3 assessments at 6-week intervals. Clinical assessments during the trial phase will be performed every three months. This will allow measuring the progression rate before and after starting treatment (either active or placebo).

ELIGIBILITY:
Inclusion Criteria:

* Probable laboratory-supported, probable, or definite ALS, as defined by El Escorial Revised ALS diagnostic criteria at screening visit (month -3)
* Disease duration ≤ 18 months at screening visit (month -3)
* Able to perform reproducible pulmonary function tests at screening visit (month -3)
* Forced vital capacity or slow vital capacity ≥70% of normal at screening visit (month -3)
* Stable on riluzole treatment for 3 months in the lead-in period
* Signed informed consent at screening visit (month -3)

Exclusion Criteria:

* Treatment with edaravone
* Other causes of neuromuscular weakness
* Presence of other neurodegenerative diseases
* Significant cognitive impairment, clinical dementia or psychiatric illness
* Severe cardiac or pulmonary disease
* Other diseases precluding functional assessments
* Other life-threatening diseases
* Any use of non-invasive ventilation (e.g. continuous positive airway pressure, non-invasive bi-level positive airway pressure or non-invasive volume ventilation) for any portion of the day, or mechanical ventilation via tracheostomy, or on any form of oxygen supplementation
* Gastrointestinal disorder that is likely to impair absorption of study drug from the gastrointestinal tract
* Has taken any investigational study drug within 30 days or five half-lives of the prior agent, whichever is longer, prior to dosing
* Any clinically significant laboratory abnormality
* Other concurrent investigational medications
* Active peptic ulcer
* Previous surgery or infections of small intestine
* Patients unable to easily swallow the treatment pills
* Acute inflammation of the gallbladder or bile ducts
* Occurrence of frequent biliary colic, biliary infections, severe pancreatic abnormalities
* Bile duct obstruction, calcified X-ray opaque gallstones and reduced mobility of the gallbladder
* Subjects who weigh 88 lbs (40 kg) or less
* Aspartate aminotransferase or alanine aminotransferase concentrations more than 3 times the upper limit of normal
* Creatinine clearance 50 ml/min or less
* Any clinically significant neurological, haematological, autoimmune, endocrine, cardiovascular, neoplastic, renal, gastrointestinal, or other disorder that, in the Investigator's opinion, could interfere with the subject's participation in the study, place the subject at increased risk, or confound interpretation of study results
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive TUDCA or that the subject is unable or unlikely to comply with the dosing schedule or study evaluations
* The patient of reproductive potential is sexually active and is not willing to use highly effective contraception during the study and up to 90 days after the day of last dose
* The patient is pregnant or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of responder patients | 18 months
  Identification of the responder patients defined as those showing an improvement of at least 20% in the ALSFRS-R slope

SECONDARY OUTCOMES:
Survival time | 18 months
  Survival time measured by death or respiratory insufficiency
ALS disease functional rating scale - revised version (ALSFRS-R) | 18 months
  Difference in change from baseline in ALSFRS-R. Each task of the scale is rated on a five-point scale from 0 = can't do, to 4 = normal ability. Individual item scores are summed to produce a reported score ranging from 0 = worst to 48 = best.
ALS Assessment Questionnaire-40 (ALSAQ-40) | 18 months
  Difference in change from baseline in ALSAQ-40. The instrument contains 40 statements that measure five dimensions of health state: Physical Mobility (10 statements), Activities of Daily Living and Independence (10 statements), Eating and Drinking (5 statements), Communication (5 statements), Emotional Functioning (10 statements). The patient must indicate how often (Never, Rarely, Sometimes, Often, or Always) the statement have been true. Dimension scores are coded on a likert scale, ranging from 0 (best health as assessed by the scale) to 100 (worse health as assessed by the measure).
Forced Vital Capacity | 18 months
  Difference in change from baseline in Forced Vital Capacity
EuroQol 5-Dimension-5 Levels (EQ-5D-5L) scale | 18 months
  Difference in change from baseline in EQ-5D-5L scale. The EQ-5D-5L descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension has 5 levels: 1.no problems, 2.slight problems, 3.moderate problems, 4.severe problems, 5.extreme problems. The patient is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the patient health state. Numbers 1-5 have no arithmetic properties and should not be used as a cardinal score.
Medical Research Council (MRC) scale | 18 months
  Difference in change from baseline in muscle force assessed by the MRC scale. The scale rates muscle strength of 6 muscles (3 at the upper and 3 at the lower limbs), bilaterally. Each muscle is graded from 0 = no movement, to 5 = normal strength, giving a total sum-score that ranges from 0 (total paralysis) to 60 (normal strength).
Neurofilaments levels | 18 months
  Effect of TUDCA on Neurofilament levels in comparison to placebo
MMP-9 levels | 18 months
  Effect of TUDCA on MMP-9 expression in comparison to placebo
Long-term safety and tolerability | 18 months
  assessed through adverse reaction, concomitant treatment, physical examination, vital signs and routine haematology and biochemistry analyses

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Albanese, MD, Study Chair — Humanitas Mirasole SpA
Locations (25):
- Katholieke Universiteit Leuven, Leuven, Belgium
- France (4):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire Limoges, Limoges
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Regional Universitaire de Tours, Tours
- Germany (6):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Alfried Krupp Krankenhaus Rüttenscheid, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Universität Ulm, Ulm
- Trinity College Dublin, Dublin, Ireland
- Italy (6):
  - IRCCS Istituto Auxologico Italiano, Milan
  - NEuroMuscular Omnicentre. Fondazione Serena Onlus, Milan
  - AOU Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Santa Maria di Terni, Terni
  - AOU Città della Salute e della Scienza di Torino, Torino
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- United Kingdom (6):
  - The Walton Centre NHS Foundation Trust, Liverpool
  - Plymouth Hospitals NHS Trust, Plymouth
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Salford Royal NHS Foundation Trust, Salford
  - University of Sheffield, Sheffield
  - Royal Stoke University Hospital, Stoke

IPD SHARING:
Plan to Share IPD: Yes
Once the dataset has been analysed, a complete, cleaned, anonymized copy of the final data used in conducting the final analyses will be made available to be used in further studies by the research partners or by other research groups and clinicians.
  To prevent misuse and misinterpretation, relevant study metadata (such as the study protocol, case report forms, documentation providing information about the methodology and procedures used to collect the data, definition of variables and statistical code) will be shared in a data repository with a stable URL. Patient anonymity and legal compliance will be assured throughout all the steps of data transfer.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Three months after the data-entry process and final data curation
Access Criteria: Data will be made available only to qualified designated persons (methodologists, biostatisticians) from other academic institutions, on request. User registration will be required in order to access files.

REFERENCES:
- [Background] Albanese A, Ludolph AC, McDermott CJ, Corcia P, Van Damme P, Van den Berg LH, Hardiman O, Rinaldi G, Vanacore N, Dickie B; TUDCA-ALS Study Group. Tauroursodeoxycholic acid in patients with amyotrophic lateral sclerosis: The TUDCA-ALS trial protocol. Front Neurol. 2022 Sep 27;13:1009113. doi: 10.3389/fneur.2022.1009113. eCollection 2022. PMID 36237618
- [Derived] Lombardo FL, Spila Alegiani S, Mayer F, Cipriani M, Lo Giudice M, Ludolph AC, McDermott CJ, Corcia P, Van Damme P, Van den Berg LH, Hardiman O, Nicolini G, Vanacore N, Dickie B, Albanese A, Puopolo M; TUDCA-ALS Study Group. A randomized double-blind clinical trial on safety and efficacy of tauroursodeoxycholic acid (TUDCA) as add-on treatment in patients affected by amyotrophic lateral sclerosis (ALS): the statistical analysis plan of TUDCA-ALS trial. Trials. 2023 Dec 5;24(1):792. doi: 10.1186/s13063-023-07638-w. PMID 38053196
- See also: TUDCA-ALS Consortium website — http://www.tudca.eu/